CLINICAL TRIAL: NCT00748982
Title: A Single-centre, Single-blind, Randomised, Placebo-controlled Phase IIa Study to Investigate the Effect of AZD1305 Given as an Intravenous (iv) Infusion on Left Ventricular Performance in Patients With Left Ventricular Dysfunction
Brief Title: Investigate the Effect of AZD1305 on Patients With Left Ventricular Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Helen Lunde, MD, Medical Science Director, Emerging Arrhythmia and Lipids, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D3190C00013; 2008-001254-41
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Results first posted 2011-06-13 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Left Ventricle Function
Keywords: AZD1305; anti-arrhythmics; safety
MeSH Terms: interventions — tert-butyl (2-(7-(2-(4-cyano-2-fluorophenoxy)ethyl)-9-oxa-3,7-diazabicyclo(3.3.1)non3-yl)ethyl)carbamate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD1305
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1305 — iv single infusion: initial iv loading dose which will be followed by a maintenance dose given for a maximum of 90 minutes
  Arms: 1
Drug: Placebo — iv single infusion: initial iv loading dose which will be followed by a maintenance dose given for a maximum of 90 minutes
  Arms: 2

SUMMARY:
To explore if AZD1305 compromises left ventricular performance in patients with left ventricular dysfunction

ELIGIBILITY:
Inclusion Criteria:

* Male patients and postmenopausal women
* Mildly/moderately decreased heart function
* Regular heart rhythm

Exclusion Criteria:

* Potassium outside normal reference values
* Child bearing potential
* Severely decreased heart function

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lund, MD, Study Director — AstraZeneca R&D, Mölndal, Sweden; Marianne Hartford, MD, Principal Investigator — AstraZeneca, Clinical Pharmacology Unit at Sahlgrenska University Hospital, Sweden
Locations (1):
- Research Site, Gothenburg, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled 33 patients and randomised 16 patients between August 2008 and July 2009 at a Clinical Pharmacology Unit located at a University Hospital in Sweden.
Pre-assignment Details: Screening for eligibility and no significant changes in the medication for heart failure during the preceding 1 month before enrolment. In addition, patients for whom it was not possible to obtain high quality echocardiographic pictures were excluded from the study. The pre-entry visit was 30 days or less before the first dosing visit.
Groups:
- AZD1305 Dose 1 and Dose 2: AZD1305 was given as an initial intravenous (iv) loading dose during 30 min followed by a maintenance iv dose during a maximum of 90 min. The infusion was stopped when all echocardiographic measurements had been carried out. The mean total dose of AZD1305 was 30 mg (range 29-31 mg)
- Placebo Dose 1 and Dose 2: Sodium chloride was given as an initial iv loading dose during 30 min followed by a maintenance iv dose during a maximum of 90 min. The infusion was stopped when all echocardiographic measurements had been carried out
Period: Overall Study
Arm/Group | AZD1305 Dose 1 and Dose 2 | Placebo Dose 1 and Dose 2
Started | 12 | 4
Completed | 12 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1305 Dose 1 and Dose 2 | Placebo Dose 1 and Dose 2 | Total
Number analyzed (Participants) | 12 | 4 | 16
Age Continuous [Mean (Standard Deviation); unit: Years] | 5 (62) | 3 (65) | 4 (254)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 12 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Ejection Fraction (LVEF), Change From Baseline
Description: To explore if AZD1305 compromises left ventricular performance in patients with left ventricular dysfunction.
Time Frame: From the iv loading dose during 30 min and the following maintenance iv dose during a maximum of 90 min. The infusion was stopped when all echocardiographic measurements had been carried out
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | AZD1305 Dose 1 and Dose 2 | Placebo Dose 1 and Dose 2
Number analyzed (Participants) | 11 | 4
Percent change | 2.00 (-0.60) [-0.60 to 4.60] | -3.25 (-6.53) [-6.53 to 0.03]

2. Secondary Outcome: Number of Subjects With at Least One Reported Adverse Event During Each Study Period and in Each Dose Group
Description: To evaluate the tolerability and safety of AZD1305 given as an iv infusion to patients with left ventricular dysfunction.
Time Frame: From randomisation to last study visit (mean infusion time 1.6 hours)
Measure: Number; unit: Participants
Arm/Group | AZD1305 Dose 1 and Dose 2 | Placebo Dose 1 and Dose 2
Number analyzed (Participants) | 12 | 4
Participants | 0 | 0

3. Secondary Outcome: Area Under Curve (AUC) ( µmol*h/L) of AZD1305
Description: To evaluate the pharmacokinetics of AZD1305, given as an iv infusion, in patients with left ventricular dysfunction
Time Frame: From the iv loading dose during 30 min and the following maintenance iv dose during a maximum of 90 min.
Measure: Mean (Full Range); unit: µmol*h/L
Arm/Group | AZD1305 Dose 1 and Dose 2 | Placebo Dose 1 and Dose 2
Number analyzed (Participants) | 12 | 0
µmol*h/L | 2.04 [1.41 to 2.88] |

4. Secondary Outcome: QTcF Interval
Description: Maximum QTcF observed for each patient. QTcF is the QT interval corrected for the RR interval using the Fridericia formula
Time Frame: Up to 24 hours following start of IV dosing.
Measure: Mean (95% Confidence Interval); unit: ms
Arm/Group | AZD1305 Dose 1 and Dose 2 | Placebo Dose 1 and Dose 2
Number analyzed (Participants) | 12 | 4
ms | 446 (409) [409 to 512] | 445 (437) [437 to 459]

ADVERSE EVENTS:
Description: Each patient can experience multiple AEs
Arm/Group | AZD1305 Dose 1 and Dose 2 | Placebo Dose 1 and Dose 2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/12 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD1305 Dose 1 and Dose 2 (N=12) | Placebo Dose 1 and Dose 2 (N=4)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI was employed at AstraZeneca and had therefore to follow AZ policy.